CLINICAL TRIAL: NCT03862599
Title: Low Intensity Extracorporeal Shock-wave Therapy (Li-ESWT) in Penile Rehabilitation After Radical Prostatectomy
Brief Title: Low Intensity Shock-wave Therapy (Li-ESWT) in Penile Rehabilitation After Radical Prostatectomy
Acronym: LiST-PRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Tet Yap, Principal Investigator, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250004
Record Dates: First submitted 2018-10-10; First posted 2019-03-05 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy
Keywords: erectile dysfunction; shockwave; treatment; prostatectomy
MeSH Terms: conditions — Erectile Dysfunction | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of probe applicator at device manufacturer before ESWT use
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care + sham ESWT (Sham Comparator): Cialis and Vacuum pump + sham Extra-corporeal shockwave therapy (ESWT)
  Interventions: Device: Extra-corporeal shockwave therapy (ESWT); Other: Standard care
- Standard care + active ESWT (Active Comparator): Cialis and Vacuum pump + active Extra-corporeal shockwave therapy (ESWT)
  Interventions: Device: Extra-corporeal shockwave therapy (ESWT); Other: Standard care

INTERVENTIONS:
Device: Extra-corporeal shockwave therapy (ESWT) — low-intensity extra-corporeal shockwave therapy
Other: Standard care — Cialis and vacuum pump

SUMMARY:
Erectile dysfunction (ED) is reported in up to 85% of men who have undergone a radical prostatectomy for prostate cancer. A few small studies have recently shown that low-intensity shockwave therapy may improve sexual performance in men with ED. However, the optimal dosage and length of treatment is yet to be determined. The investigators propose a randomised trial evaluating the efficacy and safety of low-intensity shockwave therapy in men with ED following prostatectomy surgery.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is reported in up to 85% of men who have undergone a radical prostatectomy for prostate cancer. At present, this debilitating consequence of surgery is managed in a step-wise approach including oral medication, injections and in severe cases, insertion of a penile prosthesis. A few small studies have shown that low-intensity shockwave therapy may improve sexual performance in men with ED. However, the optimal dosage and length of treatment is yet to be determined. The investigators propose a randomised trial evaluating the efficacy and safety of low-intensity shockwave therapy in men with ED following prostatectomy surgery. Low-intensity shockwave therapy would be a non-invasive treatment to preserve and improve patient's sexual function.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 65
* Diagnosed with low/intermediate-risk prostate cancer:
* PSA < 20 ng/ml
* Gleason score < 8
* PCa stage =< T2b
* Baseline IIEF-ED 17-30 without erectogenic aids
* No pre-operative urinary incontinence (no usage of urinary pads)
* Sexually active
* Able to understand and complete patient questionnaires
* Consent to participate

Exclusion Criteria:

* Anatomical abnormalities in the genitalia or pelvic region
* Post-RP complications that could impact safety or effectiveness of ESWT (eg. hematoma, fistula, unresolved anastomotic leak)
* Incomplete tumor removal (positive surgical margin)
* Tumor upstaging beyond T2b
* Nerve sparing score > 5
* Previous or scheduled treatment with pelvic radiotherapy and/or androgen deprivation therapy
* Untreated hypogonadism (serum total testosterone < 300 mg/dL)
* Anti-coagulant medication, except acetylsalicyclic acid up to 100mg daily
* Any other condition that would prevent the patient from completing the study, as judged by the principle investigator

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Function | 6 months
  Measurement of average change in IIEF-ED from baseline (pre-RP) to 24 week-FU 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction 5 being the worst outcome

SECONDARY OUTCOMES:
Penile length | 12 months
  Clinical measurement of change in stretched flaccid penile length from baseline and time points to 12 months
Urinary Incontinence | 12 months
  Measurement of average change in EPIC questionnaire from baseline (pre-RP) to 24 week-FU and time points to 12 months
Adverse Events | 12 months
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Tet Yap, FRCS (Urol), Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalyvianakis D, Memmos E, Mykoniatis I, Kapoteli P, Memmos D, Hatzichristou D. Low-Intensity Shockwave Therapy for Erectile Dysfunction: A Randomized Clinical Trial Comparing 2 Treatment Protocols and the Impact of Repeating Treatment. J Sex Med. 2018 Mar;15(3):334-345. doi: 10.1016/j.jsxm.2018.01.003. Epub 2018 Feb 1. PMID 29396020